CLINICAL TRIAL: NCT02281708
Title: A Multi-center Phase III Randomized Controlled Trial Comparing Between Adjuvant Chemotherapy and Observation in High Risk Patients With Completely Resected Stage Ib Lung Adenocarcinoma
Brief Title: Multicenter Randomized Controlled Trial Adjuvant Chemotherapy vs Observation in pStage Ib Lung Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sanghoon Jheon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRO
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Stage Ib Lung Carcinoma
Keywords: normogram; recurrence; adjuvant chemotherapy; disease free survival; Quality of life
MeSH Terms: conditions — Lung Neoplasms; Recurrence | interventions — Vinorelbine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low risk (No Intervention): low risk; observation
- high risk; observation group (No Intervention): high risk: observation
- high risk; adjuvant chemotherapy group (Experimental): high risk. vinorelbine plus cisplatin
  Interventions: Drug: vinorelbine plus cisplatin

INTERVENTIONS:
Drug: vinorelbine plus cisplatin — Drugs will be administered for 4 cycles, and should be administered at scheduled day +/- 3 days
  * vinorelbine 25mg/m2 IV (Day 1, 8) q 3wks cisplatin 75mg/m2 IV (Day 1) q 3wks
  Other Names: Navelbine (cisplatin) plus DDP
  Arms: high risk; adjuvant chemotherapy group

SUMMARY:
Researchers developed the nomogram which evaluate the risk of recurrence after surgical resection, and found that the stage 1 NSCLC patients with more than 104 point of nomogram showed similar recurrence rate to the recurrence rate of stage 2 NSCLC patients. Thus those stage 1 NSCLC patients at high recurrence rate are considered to show positive effect of adjuvant chemotherapy and perform the study to prove this hypothesis.

Applying the nomogram, the patient scored lower than 104 is categorized into low risk group and is to be grouped as the observation group which adjuvant chemotherapy will not be given. The high risk group patients (the nomogram scored larger than 104) are randomly divided into the treatment group and the observation group. Then, the clinical result on the recurrence between the observation group and the treatment group will be compared.

- Regimen of the adjuvant chemotherapy: The most commonly used 1st line chemotherapy regimen which is vinorelbine plus cisplatin will be admitted for 4 cycles. Also the three days before and the after the estimated day are permitted as allowance.

Intravenous administration of vinorelbine (25mg/m2), the 1st and the 8th day of the each cycle, every 3 weeks.

Intravenous administration of cisplatin (75mg/m2), the 1st day of the each cycle, every 3 weeks.

DETAILED DESCRIPTION:
Enrolled stage 1B adenocarcinoma patient will be registered for the study and be randomly allocated to the treatment group and the observation group by the stratification factor; the institution. Each group is determined to have same number of study population. This study is open labeled and follow the permuted block design. Also the patients will be allocated by randomized table provided by a statistician. If it is converted to e-CRF, randomization of the patients will be performed by the automated computer program.

Total 1012 patients will be enrolled to this study. Among 506 high risk stage 1B adenocarcinoma patients, patients will be allocated to the treatment and the observation groups, 253 patients each. Also 506 low risk stage 1B adenocarcinoma patients will be enrolled as the observation group. Because, among stage 1B patients, it was revealed that the high risk patients whose nomogram point exceeds 104 occupied about 50% in analysis.

Estimated 3 year disease free survival for the treatment group and the observation group is 66% and 54%, respectively. The 3 year disease free survival rate for the observation group was estimated based on retrospective multicenter study on 1132 stage 1 NSCLC patients, previously reported in Korea. During the 3 year of follow up duration, the withdrawal rate was presumed to be 10% because of loss of follow-up, violation of the consent and other causes. Study population enrollment is estimated as 48 months and mean follow-up duration is estimated as 24 months. Total duration of the study is set as 72 months. In this study design, the number of the high risk patients of each group is 253 and it supports 80% power of test with a two-sided alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet ALL of the following criteria in order to be eligible for this study
* Age ≥18 years and Age <80
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* The pathological stage Ib adenocarcinoma after complete resection (AJCC 7th). (Patients with adenocarcinoma in situ are excluded)
* Patients must have undergone pulmonary resection more than lobectomy (lobectomy, bilobectomy, pneumonectomy).
* Patients must have undergone either mediastinal lymph node dissection or systemic sampling.
* Tumor must be resected completely without gross or microscopic residual tumor.
* The interval between surgery for lung cancer and randomization must be no more than 8 weeks.
* The patients must be willing and sign informed consent prior to randomization.
* Patients with appropriate bone marrow function. ANC ≥1,500/uL, hemoglobin ≥9.0g/dL (can be corrected by transfusion). platelet ≥100,000/uL
* Patients with appropriate renal function Serum creatinine ≤ 1 x UNL(upper limit or normal) or Estimated creatinine clearance ≥ 45 ml/min
* Patients with appropriate liver function Serum bilirubin ≤ 1.5 x UNL, AST (SGOT) and ALT (SGPT) ≤ 3 x UNL, alkaline phosphatase ≤ 3 x UNL

Exclusion Criteria:

* Patients meeting any ONE of the following criteria are not eligible for this study.
* Other concurrent serious diseases that may interfere with planned treatment.
* Pregnant of lactation women
* Women of childbearing potential without a negative pregnant test (urine HCG), within 14 days prior to randomization or less than one year after menopause.
* Any previous systemic chemotherapy for cancer or anti-cancer immunotherapy.
* History of non-lung malignancies within the 5 years prior to study entry, except for the following: carcinoma in situ of the cervix, melanoma in situ.
* Serious cardiac illness or medical conditions including uncontrolled hypertension, myocardial infarction within 6 months, unstable angina pectoris, heart failure >NYHA grad II, or uncontrolled arrhythmia.
* Patients with sensitivity to vinorelbine or cisplatin.
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 year
  the time between the operation and the date of treatment for recurred lung cancer or suspected recurrence

SECONDARY OUTCOMES:
overall survival rate (OS) | 3 year, 5 year
  the time between the operation and death from any cause
quality-of-life (QoL) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanghoon Jheon, Ph.D., Study Director — Seoul National Univsersity Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Hung JJ, Jeng WJ, Chou TY, Hsu WH, Wu KJ, Huang BS, Wu YC. Prognostic value of the new International Association for the Study of Lung Cancer/American Thoracic Society/European Respiratory Society lung adenocarcinoma classification on death and recurrence in completely resected stage I lung adenocarcinoma. Ann Surg. 2013 Dec;258(6):1079-86. doi: 10.1097/SLA.0b013e31828920c0. PMID 23532112
- [Background] Okada M, Nakayama H, Okumura S, Daisaki H, Adachi S, Yoshimura M, Miyata Y. Multicenter analysis of high-resolution computed tomography and positron emission tomography/computed tomography findings to choose therapeutic strategies for clinical stage IA lung adenocarcinoma. J Thorac Cardiovasc Surg. 2011 Jun;141(6):1384-91. doi: 10.1016/j.jtcvs.2011.02.007. Epub 2011 Mar 25. PMID 21440264
- [Background] Kim HR, Kim DJ, Lee WW, Jheon S, Sung SW. The significance of maximum standardized uptake values in patients with stage I pulmonary adenocarcinoma. Eur J Cardiothorac Surg. 2009 Apr;35(4):712-6; discussion 716-7. doi: 10.1016/j.ejcts.2008.12.030. Epub 2009 Feb 10. PMID 19211260
- [Background] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Background] Cerfolio RJ, Bryant AS, Ohja B, Bartolucci AA. The maximum standardized uptake values on positron emission tomography of a non-small cell lung cancer predict stage, recurrence, and survival. J Thorac Cardiovasc Surg. 2005 Jul;130(1):151-9. doi: 10.1016/j.jtcvs.2004.11.007. PMID 15999056
- [Background] Ohtsuka T, Nomori H, Watanabe K, Kaji M, Naruke T, Suemasu K, Uno K. Prognostic significance of [(18)F]fluorodeoxyglucose uptake on positron emission tomography in patients with pathologic stage I lung adenocarcinoma. Cancer. 2006 Nov 15;107(10):2468-73. doi: 10.1002/cncr.22268. PMID 17036361
- [Result] Yoshizawa A, Motoi N, Riely GJ, Sima CS, Gerald WL, Kris MG, Park BJ, Rusch VW, Travis WD. Impact of proposed IASLC/ATS/ERS classification of lung adenocarcinoma: prognostic subgroups and implications for further revision of staging based on analysis of 514 stage I cases. Mod Pathol. 2011 May;24(5):653-64. doi: 10.1038/modpathol.2010.232. Epub 2011 Jan 21. PMID 21252858